CLINICAL TRIAL: NCT01992653
Title: A Phase Ib/II Study Evaluating the Safety, Tolerability and Anti-Tumor Activity of Polatuzumab Vedotin (DCDS4501A) in Combination With Rituximab or Obinutuzumab, Cyclophosphamide, Doxorubicin, and Prednisone in Patients With B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study of Polatuzumab Vedotin in Combination With Rituximab or Obinutuzumab, Cyclophosphamide, Doxorubicin, and Prednisone in Participants With B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29044; 2013-003541-42 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-25 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma, Non Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Doxorubicin; obinutuzumab; polatuzumab vedotin; Prednisolone; Prednisone; Rituximab

ARMS (8):
- Polatuzumab Vedotin (1.4mg) + G-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with G-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone
- Polatuzumab Vedotin (1.0mg) + R-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone; Drug: Rituximab
- Polatuzumab Vedotin (1.8mg) + G-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with G-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone
- Polatuzumab Vedotin (1.4mg) + R-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone; Drug: Rituximab
- Polatuzumab Vedotin (1.8mg) + R-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone; Drug: Rituximab
- Polatuzumab Vedotin (2.4mg) + R-CHP (Experimental): Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone; Drug: Rituximab
- Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP (Experimental): Dose Expansion: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone; Drug: Rituximab
- Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP (Experimental): Dose Expansion: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with G-CHP.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Prednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 750 milligrams per square meter (mg/m^2) IV every 3 weeks (starting from Cycle 1 Day 1), for 6 or 8 cycles.
Drug: Doxorubicin — Doxorubicin will be administered at 50 mg/m^2 IV every 3 weeks (starting from Cycle 1 Day 1), for 6 or 8 cycles.
Drug: Obinutuzumab — Obinutuzumab will be administered at 1000 milligrams (mg) IV on Cycle 1 Days 1, 8, and 15 and on Day 1 of Cycles 3-8.
  Other Names: Gazyva/Gazyvaro
  Arms: Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP; Polatuzumab Vedotin (1.4mg) + G-CHP; Polatuzumab Vedotin (1.8mg) + G-CHP
Drug: Polatuzumab Vedotin — Polatuzumab vedotin will be administered at escalating doses (at a starting dose of 1 mg/kg) IV every 3 weeks, for 6 or 8 cycles.
  Other Names: DCDS4501A
Drug: Prednisolone — Prednisolone will be administered at 100 mg orally daily for 5 days every 3 weeks (starting from Cycle 1 Day 1), for 6 or 8 cycles. Prednisone at 100 mg orally from Day -7 to Day -1 may be given at the discretion of the treating investigator physician.
Drug: Prednisone — Prednisone will be administered at 100 mg orally daily for 5 days every 3 weeks (starting from Cycle 1 Day 1), for 6 or 8 cycles. Prednisone at 100 mg orally from Day -7 to Day -1 may be given at the discretion of the treating investigator physician.
Drug: Rituximab — Rituximab will be administered at 375 mg/m^2 IV every 3 weeks (starting from Cycle 1 Day 1), for 6 or 8 cycles.
  Other Names: MabThera/Rituxan
  Arms: Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP; Polatuzumab Vedotin (1.0mg) + R-CHP; Polatuzumab Vedotin (1.4mg) + R-CHP; Polatuzumab Vedotin (1.8mg) + R-CHP; Polatuzumab Vedotin (2.4mg) + R-CHP

SUMMARY:
This multicenter, open-label, dose-escalation study will evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of polatuzumab vedotin in combination with rituximab or obinutuzumab, cyclophosphamide, doxorubicin, and prednisone (CHP chemotherapy) in participants with non-Hodgkin's lymphoma (NHL). Participants will receive escalating doses of polatuzumab vedotin intravenously (IV) every 3 weeks in combination with standard doses of rituximab plus CHP chemotherapy (R-CHP) or obinutuzumab plus CHP chemotherapy (G-CHP). Participants will be treated for a total of six or eight cycles in accordance with local institutional practice. Two parallel treatment arms will explore doses of polatuzumab vedotin in combination with R-CHP or G-CHP. The maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of polatuzumab vedotin in combination with R-CHP will be identified before it is combined with G-CHP. Once the MTD or RP2D is determined, polatuzumab vedotin will be dosed at MTD or RP2D -1 in combination with G-CHP to start the dose escalation of this combination.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* At least one bi-dimensionally measurable lesion, defined as greater than (>) 1.5 centimeters (cm) in its longest dimension
* Life expectancy of at least 24 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate hematologic function (unless inadequate function is due to underlying disease, as established by extensive bone marrow involvement or is due to hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator)
* Agreement to use highly effective contraception measures. Women of childbearing potential must agree to remain abstinent or use contraceptive measures that result in a failure rate of <1 percent (%) per year during the treatment period and for at least 12 months for R-CHP arm or for at least 18 months for G-CHP arm after the last dose of study drug. Men must agree to remain abstinent or to use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 5 months after the last dose of study drug

Dose-Escalation Portion of the Study:

* Histologically confirmed B-cell NHL: Participants with newly diagnosed B-cell NHL or relapsed/refractory B-cell NHL are eligible
* No more than one prior systemic treatment regimen for B-cell NHL (single agent anti-cluster of differentiation [CD] 20 monoclonal antibody therapy will not be counted as a prior treatment regimen)
* No prior treatment with anthracyclines

Expansion Portion of the Study:

* Previously untreated participants with diffuse large B-cell lymphoma (DLBCL)
* International Prognostic Index (IPI) score of 2-5

Exclusion Criteria:

Dose-Escalation Portion of the Study:

* Diagnosis of primary mediastinal DLBCL

Expansion Portion of the Study:

* Participants with transformed lymphoma
* Prior therapy for NHL

All Participants:

* Prior stem cell transplant
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to receive any of the individual components of R-CHP or G-CHP
* Current Grade greater than (>) 1 peripheral neuropathy
* Ongoing corticosteroid use of >30 milligrams per day (mg/day) of prednisone/prednisolone or equivalent. Participants receiving corticosteroid treatment with less than or equal to (</=) 30 mg/day of prednisone/prednisolone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration before Cycle 1 Day 1
* Primary central nervous system (CNS) lymphoma
* Vaccination with live vaccines within 6 months before Cycle 1 Day 1
* History of other malignancy that could affect compliance with the protocol or interpretation of results. Participants with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix are eligible. Participants with a malignancy that has been treated with surgery alone with curative intent will also be excluded unless the malignancy has been in documented remission without treatment for greater than or equal to (</=) 5 years before enrollment
* Evidence of significant, uncontrolled concomitant diseases, including renal disease that would preclude chemotherapy administration, or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks before Cycle 1 Day 1
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Positive for hepatitis B or hepatitis C infection
* Prior radiotherapy to the mediastinal/pericardial region
* Pregnant or lactating women
* Recent major surgery within 6 weeks before the start of Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-11-29 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (11):
- United States (7):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Washington University; Pediatrics, St Louis, Missouri
  - Northwest Cancer Specialists, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Willamette Valley Clinical Studies; Cancer Institute, Springfield, Oregon
  - Blue Ridge Cancer Care, Roanoke, Virginia
- France (4):
  - Hopital Henri Mondor, Unite Hemopathies lymphoides, Créteil
  - Hopital Claude Huriez - CHU Lille; Service des maladies du sang, Lille
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
  - Centre Henri Becquerel; Hematologie, Rouen

REFERENCES:
- [Derived] Shi R, Lu T, Ku G, Ding H, Saito T, Gibiansky L, Agarwal P, Li X, Jin JY, Girish S, Miles D, Li C, Lu D. Asian race and origin have no clinically meaningful effects on polatuzumab vedotin pharmacokinetics in patients with relapsed/refractory B-cell non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2020 Sep;86(3):347-359. doi: 10.1007/s00280-020-04119-8. Epub 2020 Aug 8. PMID 32770353
- [Derived] Tilly H, Morschhauser F, Bartlett NL, Mehta A, Salles G, Haioun C, Munoz J, Chen AI, Kolibaba K, Lu D, Yan M, Penuel E, Hirata J, Lee C, Sharman JP. Polatuzumab vedotin in combination with immunochemotherapy in patients with previously untreated diffuse large B-cell lymphoma: an open-label, non-randomised, phase 1b-2 study. Lancet Oncol. 2019 Jul;20(7):998-1010. doi: 10.1016/S1470-2045(19)30091-9. Epub 2019 May 14. PMID 31101489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 centers in 2 countries.
Pre-assignment Details: A total of 85 participants were enrolled at 11 centers in the following countries: France (31 participants) and United States (54 participants). 3 participants did not receive any study treatment (2 had exclusionary lab values and 1 withdrew) meaning that the safety population consisted of 82 participants.
Groups:
- Polatuzumab Vedotin (2.4mg) + R-CHP: Dose Escalation: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP. The participant in this group was incorrectly dosed on 2.4mg Pola R-CHP group and should have been assigned to the 1.8mg Pola R-CHP group.
- Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP: Dose Expansion: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with R-CHP. Participants treated with MTD determined from dose escalation cohorts.
- Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP: Dose Expansion: Participants will receive a total of six to eight 21-day cycles of polatuzumab vedotin in combination with G-CHP. Participants treated with MTD determined from dose escalation cohorts.
Period: Overall Study
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Started | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
Completed | 3 | 3 | 5 | 1 | 5 | 6 | 32 | 13
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 8 | 4
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP | Total
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (6.4) | 65.0 (7.0) | 67.3 (3.5) | 68.0 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 70.7 (4.5) | 60.0 (14.3) | 69.6 (7.2) | 61.6 (14.6) | 66.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 4 | 0 | 2 | 4 | 20 | 6 | 39
  Male | 3 | 0 | 2 | 1 | 4 | 2 | 20 | 11 | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 3 | 3 | 6 | 1 | 6 | 6 | 27 | 14 | 66
  Not Stated | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 12
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 5
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  White | 3 | 3 | 6 | 1 | 5 | 6 | 33 | 15 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events in Diffuse Large B-Cell Lymphoma (DLBCL) Population
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the national cancer institute common terminology criteria for AEs, Version 4.0 (NCI-CTCAE, v4.0). Reported are the number of subjects with AEs, Grade 3-5 AEs, and Serious Adverse Events (SAEs).
Time Frame: Baseline up to 5 years
Population: The safety population was defined as all participants who have received at least one dose of study medication. Results were reported for participants with DLBCL.
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Participants | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17

2. Primary Outcome: Number of Participants With Adverse Events in Non-DLBCL Population
Description: as for outcome 1
Time Frame: Baseline up to 5 years
Population: The safety population was defined as all participants who have received at least one dose of study medication. Results were reported for participants with Non-DLBCL.
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Participants | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in DLBCL Population
Description: All dose-escalation cohorts will consist of at least 3 participants. If a DLT is observed in 1 participant at a given dose level during the DLT observation period before dose escalation, additional participants will be enrolled at that dose level for a total of at least 6 participants. DLT assessment forms part of determining the Maximum Tolerated Dose (MTD). The highest dose level resulting in DLTs in less than one-third of a minimum of 6 participants will be declared the MTD.
Time Frame: Cycle (Cy) 1 Day 1 (D1) to Cy 2 D1 (cycle length=21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 0 | 0
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With DLTs in Non-DLBCL Population
Description: as for outcome 3
Time Frame: Cycle (Cy) 1 Day 1 (D1) to Cy 2 D1 (cycle length=21 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Objective Response (CR or Partial Response [PR]), as Assessed by Investigator Using Cheson Criteria for DLBCL Population
Description: Complete Response (CR) rate was defined as the percentage of participants with CR at the end of treatment, as assessed by the investigator, with and without FDG-PET. The overall response rate was defined as the percentage of participants with CR or PR at the end of treatment, as assessed by the investigator, with and without FDG-PET.
Time Frame: At the end of treatment (Month 6)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Percentage of Participants
  Complete Response (CR) | 50.0 [2.53 to 97.47] | 100.0 [36.84 to 100.00] | 100.0 [54.93 to 100.00] |  | 75.0 [24.86 to 98.73] | 100.0 [47.29 to 100.0] | 75.0 [61.29 to 85.76] | 76.5 [53.95 to 91.54]
  Partial Response (PR) | 50.0 [2.53 to 97.47] | 0 [0.00 to 63.16] | 0 [0.00 to 45.07] |  | 0 [0.00 to 52.71] | 0 [0.00 to 52.71] | 15.0 [6.74 to 27.47] | 11.8 [2.13 to 32.62]

6. Secondary Outcome: Percentage of Participants With Objective Response (CR or Partial Response [PR]), as Assessed by Investigator Using Cheson Criteria for Non-DLBCL Population
Description: as for outcome 5
Time Frame: At the end of treatment (Month 6)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Percentage of Participants
  Complete Response (CR) | 100.0 [5.00 to 100.00] |  | 100.0 [5.00 to 100.00] | 100.0 [5.00 to 100.00] | 100.0 [22.36 to 100.00] | 100.0 [22.36 to 100.0] |  |
  Partial Response (PR) | 0 [0.00 to 95.00] |  | 0 [0.00 to 95.00] | 0 [0.00 to 95.00] | 0 [0.00 to 77.64] | 0 [0.00 to 77.64] |  |

7. Secondary Outcome: Number of Participants With Anti-Polatuzumab Vedotin Antibodies
Description: The Anti-Drug Antibody (ADA) screening assay was optimized to tolerate drug interference and was able to detect 90 and 500 ng/mL of the positive control sample in the presence of 20 μg/mL of polatuzumab vedotin. Polatuzumab vedotin total antibody concentrations were determined for each ADA sample. Out of a total of 186 ADA samples that were measured for polatuzumab vedotin total antibody, 184 samples had levels less than 20 μg/mL. Polatuzumab vedotin total antibody concentrations ranged from <0.050 μg/mL to 52.1 μg/mL with a median concentration of 3.38 μg/mL.
Time Frame: Baseline up to Month 9 (assessed prior to polatuzumab vedotin infusion [0 hour; Hr] on Day 2 [D2] of Cy 1 and 2, D1 of Cy 4, treatment completion/early termination [Month 6], and at 3 months post-treatment [Month 9]; cycle length=21 days)
Population: The safety population was defined as all participants who have received at least one dose of study medication. Results were reported for participants with DLBCL and Non-DLBCL.
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Anti-Obinutuzumab Antibodies
Description: The ADA screening assay was optimized to tolerate drug interference and was able to detect 500 ng/mL of the ADA-positive control sample in the presence of 50 micrograms/mL of obinutuzumab. Obinutuzumab concentrations were determined for each ADA sample. Out of a total of 48 ADA samples that were measured for obinutuzumab, 9 samples had levels less than 50 micrograms/mL of obinutuzumab. Obinutuzumab concentrations in ADA samples ranged from 0.282 micrograms/mL to 522 micrograms/mL with a median concentration of 210 micrograms/mL. Therefore, it is possible that samples with obinutuzumab concentrations greater than 50 micrograms/mL might be false negative for ADA.
Time Frame: Baseline up to Month 9 (assessed prior to obinutuzumab infusion [0 Hr] on D1 of Cy 1, 2, 4 and at 3 months post-treatment [Month 9]; cycle length=21 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Polatuzumab Vedotin
Description: AUC information for Polatuzumab Vedotin was estimated from serum concentration data using non-compartmental analysis.
Time Frame: Pre-polatuzumab vedotin infusion (Hr 0), 30 minutes (min) post-infusion (infusion time=30-90 min) on D 2 of Cy 1, 2 & D1 of Cy 3, 4; Cy 1 Days 8 & 15; Cy 3 Day 8; at end of treatment (Month 6), at Month 3 follow-up (Month 9) (cycle length=21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng day/mL
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
ng day/mL | 1300 (22) | 1510 (354) | 2600 (413) | 4090 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 1940 (154) | 1850 (491) | 1870 (527) | 1940 (482)

10. Secondary Outcome: Maximum Concentration (Cmax) of Polatuzumab Vedotin
Description: Cmax for Polatuzumab Vedotin was estimated from serum concentration data using non-compartmental analysis.
Time Frame: Pre-polatuzumab vedotin infusion (Hr 0), 30 min post-infusion (infusion time=30-90 min) on D 2 of Cy 1, 2 & D1 of Cy 3, 4; Cy 1 Days 8 & 15; Cy 3 Day 8; at end of treatment (Month 6), at Month 3 follow-up (Month 9) (cycle length=21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
ng/mL | 373 (147) | 537 (184) | 781 (72.6) | 1400 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 537 (59.1) | 557 (114) | 532 (163) | 530 (138)

11. Secondary Outcome: Clearance (CL) of Polatuzumab Vedotin
Description: CL for Polatuzumab Vedotin was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
mL/day/kg | 14.0 (0.370) | 17.3 (4.16) | 12.8 (2.05) | 10.5 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 13.2 (1.29) | 18.7 (5.30) | 18.9 (5.27) | 17.7 (3.83)

12. Secondary Outcome: Terminal Half-Life (t1/2) of Polatuzumab Vedotin
Description: t1/2 for Polatuzumab Vedotin was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
days | 5.03 (0.905) | 4.85 (0.720) | 4.79 (0.675) | 4.42 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 5.19 (0.430) | 4.89 (0.526) | 5.03 (0.621) | 5.50 (0.795)

13. Secondary Outcome: Steady-State Volume of Distribution (Vss) of Polatuzumab Vedotin
Description: Vss for Polatuzumab Vedotin was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 6 | 40 | 17
mL/kg | 58.2 (9.92) | 80.0 (9.97) | 57.7 (7.95) | 41.9 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 67.9 (7.42) | 87.5 (19.3) | 96.5 (34.1) | 99.3 (27.4)

14. Secondary Outcome: Plasma Levels of Cyclophosphamide
Description: Plasma levels of cyclophosphamide will be assessed and compared at the same timepoints of Cycle 1 (in the absence of polatuzumab vedotin) and Cycle 3 (in the presence of polatuzumab vedotin), and compared with historical data to evaluate potential PK interactions with polatuzumab vedotin.
Time Frame: End of cyclophosphamide infusion (infusion time=1-24 Hr), 3 and 23 hours post end of cyclophosphamide infusion on D1 of Cy 1 and 3 (cycle length=21 days)
Population: The safety population was defined as all participants who have received at least one dose of study medication. Plasma levels of cyclophosphamide were only assessed in the 'Expansion' cohorts and only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 17
ug/mL
  C1D1 0.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 13
  C1D1 0.5hr POSTDOSE |  |  |  |  |  |  | 37.5 (24.4) | 32.3 (7.64)
  C1D1 3.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 13
  C1D1 3.5hr POSTDOSE |  |  |  |  |  |  | 23.2 (2.38) | 22.5 (3.69)
  C1D1 23.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 14
  C1D1 23.5hr POSTDOSE |  |  |  |  |  |  | 2.98 (1.39) | 3.32 (1.50)
  C3D1 0.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 15
  C3D1 0.5hr POSTDOSE |  |  |  |  |  |  | 34.8 (6.14) | 35.2 (13.4)
  C3D1 3.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 16
  C3D1 3.5hr POSTDOSE |  |  |  |  |  |  | 24.2 (3.87) | 22.5 (4.26)
  C3D1 23.5hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 14
  C3D1 23.5hr POSTDOSE |  |  |  |  |  |  | 3.17 (1.66) | 3.16 (1.68)

15. Secondary Outcome: Plasma Levels of Doxorubicin
Description: Plasma levels of doxorubicin will be assessed and compared at the same timepoints of Cycle 1 (in the absence of polatuzumab vedotin) and Cycle 3 (in the presence of polatuzumab vedotin), and compared with historical data to evaluate potential PK interactions with polatuzumab vedotin.
Time Frame: 2, 24 hours post end of doxorubicin infusion (infusion time=15 min) on D1 of Cy 1 and 3 (cycle length=21 days)
Population: The safety population was defined as all participants who have received at least one dose of study medication. Plasma levels of doxorubicin were only assessed in the 'Expansion' cohorts and only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 17
ug/mL
  C1D1 2hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 11
  C1D1 2hr POSTDOSE |  |  |  |  |  |  | 35.4 (13.6) | 30.2 (6.82)
  C1D1 24hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 12
  C1D1 24hr POSTDOSE |  |  |  |  |  |  | 9.13 (2.51) | 11.7 (11.6)
  C3D1 2hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 16
  C3D1 2hr POSTDOSE |  |  |  |  |  |  | 29.3 (10.9) | 29.6 (10.8)
  C3D1 24hr POSTDOSE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 14
  C3D1 24hr POSTDOSE |  |  |  |  |  |  | 8.68 (2.05) | 9.14 (2.12)

16. Secondary Outcome: Peripheral Neuropathy Symptom Severity: Therapy-Induced Neuropathy Assessment Scale (TINAS) Overall Neuropathy Severity Score
Description: The TINAS is an 11-item questionnaire scored on a 0 to 10 scale, with 0 being the symptom is not present to 10 being the symptom is as bad as the participant can imagine. The questionnaire will be analyzed for the individual neuropathy symptoms experienced by a participant as well as the calculation of an overall neuropathy severity score. The TINAS scale will be completed daily over the course of study treatment. Additionally, to collect information about the reversibility of peripheral neuropathy, the TINAS will be completed once a week for the first 2 months, then once a month for the next 10 months following treatment completion. Results are only being reported here up until the End of Treatment visit (duration of Study treatment).
Time Frame: Weekly up to Month 6 (22 weeks). TINAS data were collected daily, though for the analysis purpose for each participant, only the first record of each week was selected.
Population: The safety population was defined as all participants who have received at least one dose of study medication. TINAS was only assessed in the 'Expansion' cohorts and only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: Score of a Questionnaire
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 17
Score of a Questionnaire
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Baseline |  |  |  |  |  |  | 0 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 0.32 (0.45)
  Week 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Week 1 |  |  |  |  |  |  | 0 (0) | 0.91 (0.92)
  Week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  Week 2 |  |  |  |  |  |  | 0.02 (0.04) | 0.07 (0.16)
  Week 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
  Week 3 |  |  |  |  |  |  | 0.06 (0.10) | 0.22 (0.44)
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
  Week 4 |  |  |  |  |  |  | 0.18 (0.36) | 0.26 (0.63)
  Week 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
  Week 5 |  |  |  |  |  |  | 0.16 (0.32) | 0.17 (0.41)
  Week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Week 6 |  |  |  |  |  |  | 0.16 (0.32) | 0.25 (0.57)
  Week 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Week 7 |  |  |  |  |  |  | 0.14 (0.28) | 0.35 (0.77)
  Week 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8
  Week 8 |  |  |  |  |  |  | 0.17 (0.37) | 0.31 (0.59)
  Week 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8
  Week 9 |  |  |  |  |  |  | 0.25 (0.47) | 0.38 (0.61)
  Week 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 10 |  |  |  |  |  |  | 0.30 (0.41) | 0.53 (0.71)
  Week 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 11 |  |  |  |  |  |  | 0.26 (0.35) | 0.39 (0.73)
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 12 |  |  |  |  |  |  | 0.30 (0.43) | 0.65 (1.02)
  Week 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 8
  Week 13 |  |  |  |  |  |  | 0.25 (0.32) | 0.78 (1.34)
  Week 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Week 14 |  |  |  |  |  |  | 0.49 (0.86) | 0.62 (1.05)
  Week 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Week 15 |  |  |  |  |  |  | 0.48 (0.86) | 0.70 (1.28)
  Week 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8
  Week 16 |  |  |  |  |  |  | 0.66 (0.94) | 1.12 (1.61)
  Week 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7
  Week 17 |  |  |  |  |  |  | 0.25 (0.52) | 0.91 (1.44)
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 18 |  |  |  |  |  |  |  | 0.64 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.
  Week 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 19 |  |  |  |  |  |  |  | 0.45 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.
  Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 22 |  |  |  |  |  |  |  | 0.09 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.

17. Secondary Outcome: Peripheral Neuropathy Symptom Interference: TINAS Numbness/Tingling Item Score
Description: The TINAS is an 11-item questionnaire scored on a 0 to 10 scale, with 0 being the symptom is not present to 10 being the symptom is as bad as the patient can imagine. The questionnaire will be analyzed for the individual neuropathy symptoms experienced by a participant as well as the calculation of an overall neuropathy severity score. The TINAS scale will be completed daily over the course of study treatment. Additionally, to collect information about the reversibility of peripheral neuropathy, the TINAS will be completed once a week for the first 2 months, then once a month for the next 10 months following treatment completion. Additionally, a single item that asks patients to rate when numbness and tingling was at the worst will be used to predict the onset of peripheral neuropathy. The measure takes less than 5 minutes to complete. Results are only being reported here up until the End of Treatment visit (duration of Study treatment).
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score of a Questionnaire
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 17
Score of a Questionnaire
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Baseline |  |  |  |  |  |  | 0 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated. | 0 (0)
  Week 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Week 1 |  |  |  |  |  |  | 0 (0) | 1 (1.73)
  Week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  Week 2 |  |  |  |  |  |  | 0.25 (0.50) | 0 (0)
  Week 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
  Week 3 |  |  |  |  |  |  | 0.33 (0.58) | 0.40 (0.89)
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
  Week 4 |  |  |  |  |  |  | 0.40 (0.55) | 0.50 (1.22)
  Week 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
  Week 5 |  |  |  |  |  |  | 0.40 (0.55) | 0.17 (0.41)
  Week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Week 6 |  |  |  |  |  |  | 0.40 (0.55) | 0.40 (0.89)
  Week 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Week 7 |  |  |  |  |  |  | 0.29 (0.49) | 0.60 (1.34)
  Week 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8
  Week 8 |  |  |  |  |  |  | 0.33 (0.52) | 0.25 (0.71)
  Week 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8
  Week 9 |  |  |  |  |  |  | 0.40 (0.55) | 0.50 (1.07)
  Week 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 10 |  |  |  |  |  |  | 0.86 (1.21) | 1.14 (1.46)
  Week 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 11 |  |  |  |  |  |  | 0.86 (1.21) | 0.57 (1.13)
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Week 12 |  |  |  |  |  |  | 1.14 (1.21) | 0.71 (1.25)
  Week 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 8
  Week 13 |  |  |  |  |  |  | 0.86 (1.21) | 1.12 (1.81)
  Week 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Week 14 |  |  |  |  |  |  | 1.12 (1.73) | 0.88 (1.36)
  Week 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Week 15 |  |  |  |  |  |  | 1.12 (1.73) | 0.75 (1.16)
  Week 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8
  Week 16 |  |  |  |  |  |  | 1.56 (2.07) | 1.50 (1.69)
  Week 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7
  Week 17 |  |  |  |  |  |  | 0.40 (0.55) | 1.14 (1.46)
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 18 |  |  |  |  |  |  |  | 2 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.
  Week 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 19 |  |  |  |  |  |  |  | 2 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.
  Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 22 |  |  |  |  |  |  |  | 1 (NA) — Due to there being only 1 participant in this group, the SD could not be estimated.

18. Secondary Outcome: Duration of Response, as Assessed by Investigator Using Cheson Criteria for DLBCL Population
Description: Time from the date of the first occurrence of a documented CR or PR to the date of disease progression, relapse or death from any cause (PFS), as assessed by the investigator for the subgroup of participants with a best overall response of CR or PR. For participants achieving a response who did not experience disease progression, relapse, or died prior to the time of the analysis, the DOR was censored on the date of last disease assessment.
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [14.03 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [27.93 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest.

19. Secondary Outcome: Duration of Response, as Assessed by Investigator Using Cheson Criteria for Non-DLBCL Population
Description: as for outcome 18
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | 4.11 [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  |

20. Secondary Outcome: Progression Free Survival, as Assessed by Investigator Using Cheson Criteria for DLBCL Population
Description: Time from date of first dose of study drug (Day 1) to the first occurrence of progression or relapse, or death from any cause while in the study, as assessed by the investigator. If a participant did not experience progressive disease or death, PFS was censored on the day of the last tumor assessment. If a post-baseline assessment was not available, PFS was censored on Day 1.
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [17.02 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | NA [7.79 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [30.62 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest.

21. Secondary Outcome: Progression Free Survival, as Assessed by Investigator Using Cheson Criteria for Non-DLBCL Population
Description: as for outcome 20
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | 6.87 [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  |

22. Secondary Outcome: Event Free Survival, as Assessed by Investigator Using Cheson Criteria for DLBCL Population
Description: Time from randomization to disease progression or relapse, as assessed by the investigator, death from any cause, or initiation of any new anti-lymphoma therapy (NALT). If the specified event (disease progression or relapse, death, initiation of a NALT) did not occur, EFS was censored at the date of last tumor assessment. For participants without an event who did not have post-baseline tumor assessments, EFS was censored at the time of randomization.
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [17.02 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | NA [3.42 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [5.88 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | 35.45 [28.32 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest.

23. Secondary Outcome: Event Free Survival, as Assessed by Investigator Using Cheson Criteria for Non-DLBCL Population
Description: as for outcome 22
Time Frame: Screening up to disease progression or death, whichever occurs first (up to approximately 2.75 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | 6.87 [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | 6.70 [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  |

24. Secondary Outcome: Relative Dose Intensity of Polatuzumab Vedotin (Ratio of the Amount of Drug Actually Administered to the Amount Planned) for DLBCL Population
Description: Relative dose intensity (DI) was defined as the ratio of the amount of a drug actually administered (actual DI) to the amount planned (planned DI) for a fixed time period, expressed as a percentage.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Percentage | 100.70 (0.99) | 99.97 (0.55) | 96.04 (4.81) |  | 99.35 (3.19) | 99.95 (0.75) | 96.71 (6.99) | 98.92 (3.74)

25. Secondary Outcome: Relative Dose Intensity of Polatuzumab Vedotin (Ratio of the Amount of Drug Actually Administered to the Amount Planned) for Non-DLBCL Population
Description: as for outcome 24
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Percentage | 100.00 (NA) — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | 100.94 (NA) — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | 132.22 (NA) — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | 99.72 (0.06) | 100.17 (0.14) |  |

26. Secondary Outcome: Overall Survival for DLBCL Population
Description: The time from the date of randomization to the date of death from any cause. For participants who did not die at the time of the analyses, OS was censored on the last date when the participants were known to be alive.
Time Frame: Screening up to death due to any cause (up to approximately 6 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 2 | 3 | 5 | 0 | 4 | 4 | 40 | 17
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | NA [7.79 to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest.

27. Secondary Outcome: Overall Survival for Non-DLBCL Population
Description: as for outcome 26
Time Frame: Screening up to death due to any cause (up to approximately 6 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Months | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  | 15.24 [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. | NA [NA to NA] — Median, Lower and Upper Limit could not be estimated because very few participants had the event of interest. |  |

ADVERSE EVENTS:
Time Frame: 5 years
Description: The safety population was defined as all participants who received at least one dose of study medication. AEs that were entered into the data base at the time of the data base lock were included in the AE analysis.
Arm/Group | Polatuzumab Vedotin (1.0mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + R-CHP | Polatuzumab Vedotin (1.8mg) + R-CHP | Polatuzumab Vedotin (2.4mg) + R-CHP | Polatuzumab Vedotin (1.4mg) + G-CHP | Polatuzumab Vedotin (1.8mg) + G-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 0/1 | 1/6 | 0/6 | 4/40 | 2/17
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 4/6 | 0/1 | 1/6 | 3/6 | 15/40 | 6/17
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 1/1 | 6/6 | 6/6 | 40/40 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polatuzumab Vedotin (1.0mg) + R-CHP (N=3) | Polatuzumab Vedotin (1.4mg) + R-CHP (N=3) | Polatuzumab Vedotin (1.8mg) + R-CHP (N=6) | Polatuzumab Vedotin (2.4mg) + R-CHP (N=1) | Polatuzumab Vedotin (1.4mg) + G-CHP (N=6) | Polatuzumab Vedotin (1.8mg) + G-CHP (N=6) | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP (N=40) | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP (N=17)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 4 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polatuzumab Vedotin (1.0mg) + R-CHP (N=3) | Polatuzumab Vedotin (1.4mg) + R-CHP (N=3) | Polatuzumab Vedotin (1.8mg) + R-CHP (N=6) | Polatuzumab Vedotin (2.4mg) + R-CHP (N=1) | Polatuzumab Vedotin (1.4mg) + G-CHP (N=6) | Polatuzumab Vedotin (1.8mg) + G-CHP (N=6) | Expansion: Polatuzumab Vedotin (1.8mg) + R-CHP (N=40) | Expansion: Polatuzumab Vedotin (1.8mg) + G-CHP (N=17)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (5) | 14 (24) | 3 (7)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 3 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (16) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (8) | 0 (0) | 3 (3) | 5 (5) | 13 (22) | 6 (9)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (2) | 6 (16) | 6 (6)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EXCESSIVE CERUMEN PRODUCTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AMBLYOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 11 (14) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7) | 1 (1) | 2 (4) | 2 (2) | 17 (25) | 11 (14)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (5) | 4 (7) | 1 (1) | 3 (3) | 3 (3) | 16 (26) | 10 (12)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 3 (4)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (12) | 1 (4)
CATHETER SITE PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
DEVICE RELATED THROMBOSIS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
FATIGUE (General disorders) | 2 (2) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 16 (29) | 11 (16)
FEELING HOT (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILL-DEFINED DISORDER (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 9 (11) | 4 (4)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 2 (2)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD LACTIC ACID INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STREPTOCOCCUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 5 (6)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 2 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 1 (2)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 4 (5)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (5)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
DYSTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPOGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 2 (3) | 2 (3) | 5 (7) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (4)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
AFFECT LABILITY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NIGHTMARE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINE FLOW DECREASED (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR OEDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (3)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (5) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 4 (4) | 4 (7) | 4 (5)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (16) | 1 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT01992653/Prot_SAP_000.pdf